CLINICAL TRIAL: NCT05998564
Title: Comparison of the Skin Conductance Algesimeter and the Nociception Level Index in the Paediatric Population. An Observational Study.
Acronym: NOLvsSCA
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-16214
Record Dates: First submitted 2023-07-25; First posted 2023-08-21 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2023-06

CONDITIONS: Nociceptive Pain; Anesthesia; Pain
Keywords: Nociception monitoring; Pediatric population
MeSH Terms: conditions — Nociceptive Pain; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients aged 1 to 4 years of age: Patients will be connected to the NOL monitor and the SCA monitor during surgery with general anaesthesia.
  Interventions: Device: Connecting patients to both non-invasive monitors to observe and compare the monitor's capabilities.
- Patients aged 5 to 12 years of age: Patients will be connected to the NOL monitor and the SCA monitor during surgery with general anaesthesia.
  Interventions: Device: Connecting patients to both non-invasive monitors to observe and compare the monitor's capabilities.

INTERVENTIONS:
Device: Connecting patients to both non-invasive monitors to observe and compare the monitor's capabilities. — All patients will be connected to the NOL monitor and the SCA monitor during general anesthesia.

SUMMARY:
Evaluation and comparison of the skin conductance algesimeter(SCA) and the nociception level index(NOL) in the paediatric population (1-12 years) during surgery with general anaesthesia with bispectral index(BIS) in a tertiary hospital in The Netherlands.

DETAILED DESCRIPTION:
Intraoperative non-invasive monitors designed to detect nociception during surgery have seen a considerable development over the past few years. There are multiple commercial monitoring devices available of which most have not been extensively evaluated in the pediatric population. Adequate levels of perioperative analgesia are important as they lead to less intraoperative nociception and less post-operative pain and post-operative complications and thereby leads to improved patient recovery. Monitoring the nociceptive state of a patient by monitoring the autonomic peripheral sympathetic pathways during surgery with these monitoring methods might lead to earlier detection of nociception and therefore less nociception and perioperative pain. Most monitoring devices have not been extensively evaluated in the pediatric population and have not yet demonstrated large clinical implications such as a decrease in post-operative pain or a decrease in opioid usage by using monitor guided analgesia administration. One of the nociception monitoring methods that has not been studied extensively in the pediatric population is the Nociception level index(NOL, Medasense, Ramat Gan, Israel). This monitor is a multi-parametric non-invasive monitoring method that measures heartrate, heartrate variability, skin temperature, photoplethysmographic amplitude, skin conductance and fluctuations in skin conductance using a non-invasive finger probe. These parameters are combined in an algorithm that provides an index from 0-100 with an abstract unit. With 0 indicating no nociception and 100 indicating severe nociception. A first study in the paediatric population with the NOL monitor showed that the NOL index was able to significantly detect first incision and significantly respond to opioid administration during surgery in children 1 to 5 years of age. Another more recent study demonstrated that the NOL index can quantify nociceptive stimuli in children aged 1 to 12. Other more commonly used monitoring methods for nociception such as fluctuations in mean arterial blood pressure(MAP), heartrate(HR) and respiratory rate(RR) did not show a significant change during first incision or during opioid administration in this study, indicating that the NOL monitor might be a better method to assess and respond to intraoperative nociception than fluctuations in MAP, HR and RR alone.

Another nociception monitoring method is the skin conduction algesimeter(SCA, Medstorm, Oslo, Norway. This is a single parameter nociception monitoring device that uses three electrodes that are fixed to the skin to measure fluctuations in skin conductance in order to detect nociception. It measures the amount of bursts in the skin sympatetic nerves in peaks per second. This contrasts with the multiparametric design of the NOL monitor with an algorithm and an abstract index of 0-100. The SCA monitor system doesn't utilize heartrate and photoplethysmographic amplitude. Hypothetically making the device less susceptible to interference of intraoperative hemodynamic changes and intraoperative vasoactive medication administration in comparison with the NOL monitor which does utilizes these variables in its system and algorithm. Furthermore as the SCA monitor measures the direct burst of the palmary or plantary sympathetic nerves this could mean that it responds faster than the NOL index to nociceptive stimuli. The SCA monitor has already been studied in the unanesthetized and the sedated pediatric and neonatal population. But has not seen extensive validation during surgery under general anaesthesia. One small pilot study in the pediatric population under general anaesthesia has been performed. In this study only 12 patients were included, and these patients had a broad age range (8.4 ± 5 years) and received perioperative analgesia through means of continuous infusion of remifentanil. Furthermore the studies researchers did not use the recommended threshold value for the SCA monitor. Both monitors use different proprietary owned algorithms with the same aim of detecting nociception.

Therefore, the primary goal of this study is to evaluate the SCA in the pediatric population during general anaesthesia. As more extensive evaluation of the SCA in the pediatric population is imperative in order to assess if it the SCA can detect nociceptive stimuli during general anesthesia. Another primary objective of this study will be to compare the SCA with the NOL index during general anesthesia. Evaluation of SCA through this feasibility study and comparison with the NOL monitor at the same time, may answer the question of which monitor can better predict and monitor nociceptive stimulation in the perioperative period. This will be the basis for future interventional randomized studies to assess if perioperative monitoring of the analgesia level leads to improved post-operative outcomes. We hypothesize that the NOL monitor and SCA monitor will both be able to quantify nociceptive stimuli, and that the SCA monitor responds faster than the NOL monitor.

Another secondary aim of the current study is the comparison of the BIS to the algesimeters awakening index.

Previous studies have demonstrated that fluctuations in skin conductance with an increase of area under the skin conductance peaks curve while awakening from general anesthesia performs similar to the bispectral index (BIS) in the adult population during nociceptive stimuli.

Primary Objectives:

1. Evaluate if the SCA can detect nociceptive stimuli in children undergoing surgery with general anaesthesia.
2. Compare the response of the SCA to the response of the NOL monitor during surgery with general anaesthesia.

Secondary Objective(s):

1. Evaluate the response of the SCA and NOL to intraoperative opioid administration.
2. Evaluate the response of the SCA and NOL index to intraoperative administration of vasoactive medication.
3. Evaluate the response of the SCA and NOL to changes in mean arterial blood pressure (MAP, heartrate (HR) and respiratory rate (RR)
4. Comparison of the SCA awakening index to the BIS.
5. Comparison of the peak(maximum) values for NOL and SCA across both selected age groups (1-4 and 5-12)
6. Comparison of the reaction time of both monitors after nociceptive stimulation.
7. Compare the functionality of the NOL index and SCA monitor during general anesthesia and usage of localregional anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* ASA I, ASA II and ASA III
* Aged 1 to 12 years old
* Scheduled to undergo elective surgery with general anaesthesia
* Written informed consent obtained from subject or/and subject's legal representatives.

Exclusion Criteria:

* Known allergy to the adhesive tape used in the sensors.
* Patients that do not meet the inclusion criteria will be excluded.
* No free available limb to attach the probes to.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A total of 50 patients. 25 patients aged 1-4 years old, and 25 patients aged 5-12 years old that are scheduled to undergo elective surgery under general anaesthesia. Patients will be enrolled after obtaining written informed consent. We decided to evaluate the SCA and NOL index in two age groups because of the significant differences of maturations of the bodies across different ages that might influence the measurements made by the SCA and NOL monitor. Furthermore the maturation of the brain of a paediatric patient also differs significantly across different ages. Leading to significant differences in EEG patterns and corresponding BIS monitor values across age groups 1-4 and groups 5-11. Therefore, assessing the NOL and SCA in these two difference age groups results in a better ability to assess the homogeneity of the population as we will also be able to quantify and compare the depth of anesthesia through BIS monitor in these two age groups.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-09-29 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-10-25 (Actual)

PRIMARY OUTCOMES:
Changes in the SCA prior to and during a nociceptive event during the intraoperative period. | Through study completion, an average of 1 year
  The pre stimulation values for SCA will be estimated by taking the peak(maximum) value -30 to 0 seconds before the occurrence of the nociceptive event. Post stimulation values for SCA will be estimated by taking the peak (maximum) value +0 to +30 seconds after the nociceptive event.
  The SCA monitor records skin conductance in peaks per second. Varying from 0.00 peaks per second to 0,40 or more peaks per second. These peaks per second correlate with the pain index according to the manufacturer. With 0.00-0.06 peaks per second equalling pain index of zero and 0,40 or more peaks per second equalling a pain index of ten during surgical stimuli.
Changes in the NOL index prior to and during a nociceptive event during the intraoperative period. | Through study completion, an average of 1 year
  The pre stimulation values for NOL will be estimated by taking the peak(maximum) value -30 to 0 seconds before the occurrence of the nociceptive event. Post stimulation values for NOL will be estimated by taking the peak (maximum) value +0 to +30 seconds after the nociceptive event.
  The NOL index ranges from 0 to 100. With 0 indicating absence of nociception and 100 indicating severe nociception. The NOL index values are registered at a 5 second interval.
Correlation between changes in SCA and changes in NOL index during nociceptive events in the intraoperative period. | Through study completion, an average of 1 year
  The pre stimulation values for SCA and NOL will be estimated by taking the peak(maximum) value -30 to 0 seconds before the occurrence of the nociceptive event. Post stimulation values for NOL and SCA will be estimated by taking the peak (maximum) value +0 to +30 seconds after the nociceptive event.
  To compare the diagnostic performance of the SCA and the NOL index we will display data of the SCA and NOL index response to nociception stimuli in a scatterplot and we will perform an intraclass correlation coefficient calculation in order to assess if the response of the patients to the monitors correlate with each other.
  The NOL index ranges from 0 to 100. With 0 indicating absence of nociception and 100 indicating severe nociception.

SECONDARY OUTCOMES:
SCA response to opioid administration. | Through study completion, an average of 1 year.
  Response of the SCA to opioids administration is measured by comparing the peak (maximum) -20 to 0 seconds SCA value prior to fentanyl administration to the estimated peak (maximum) value +0-10 to 120-240 seconds after fentanyl administration. This is in accordance with known fentanyl pharmacokinetics in literature that states a maximum time to onset of 90 seconds
NOL response to opioid administration. | Through study completion, an average of 1 year.
  Response of the NOL index to opioids administration is measured by comparing the peak (maximum) -20 to 0 seconds NOL index value prior to fentanyl administration to the estimated peak (maximum) value +0-10 to 120-240 seconds after fentanyl administration. This is in accordance with known fentanyl pharmacokinetics in literature that states a maximum time to onset of 90 seconds.
SCA response to vasoactive medication administration. | Through study completion, an average of 1 year.
  The pre vasoactive medication values for SCA will be estimated by taking the peak(maximum) value -30 to 0 seconds before the occurrence of the nociceptive event. Post vasocative medication values for SCA will be estimated by taking the peak(maximum) value +0 to +30 seconds after the nociceptive event.
NOL response to vasoactive medication administration. | Through study completion, an average of 1 year.
  The pre vasoactive medication values for NOL will be estimated by taking the peak(maximum) value -30 to 0 seconds before the occurrence of the nociceptive event. Post vasocative medication values for NOL will be estimated by taking the peak(maximum) value +0 to +30 seconds after the nociceptive event.
Correlation between changes in the SCA compared to other predictors of nociception. | Through study completion, an average of 1 year.
  being heartrate, respiratory rate and non-invasive blood pressure data collected during nociceptive events. Data on non-invasive blood pressure is registered at a five-minute interval by the Intellivue Philips monitor (Koninklijke Philips N.V., 2004 - 2022). Data on respiratory rate is registered at a 1-minute interval by the Intellivue Philips monitor. Data on heartrate is registered at a 5 second interval by the PMD-200 monitor.
Correlation between changes in the NOL index compared to other predictors of nociception | Through study completion, an average of 1 year.
  being heartrate, respiratory rate and non-invasive blood pressure data collected during nociceptive events. Data on non-invasive blood pressure is registered at a five-minute interval by the Intellivue Philips monitor (Koninklijke Philips N.V., 2004 - 2022). Data on respiratory rate is registered at a 1-minute interval by the Intellivue Philips monitor. Data on heartrate is registered at a 5 second interval by the PMD-200 monitor.
BIS monitor response to intraoperative nociceptive stimuli | Through study completion, an average of 1 year.
  During intra-operative nociceptive events SCA awakening index and BIS will be compared in order to assess their similarity when assessing awakening from nociceptive stimuli. Appropriate statistical analysis will be performed according to the distribution of data regarding BIS and SCA awakening index.
  BIS values range from 0 to 100. A value of 0 represents the absence of brain activity, and 100 represents the awake state.
SCA awakening index response to intraoperative nociceptive stimuli | Through study completion, an average of 1 year.
  During intra-operative nociceptive events SCA awakening index and BIS will be compared in order to assess their similarity when assessing awakening from nociceptive stimuli. Appropriate statistical analysis will be performed according to the distribution of data regarding BIS and SCA awakening index.
Peak values for NOL and SCA for age group 1-4 years | Through study completion, an average of 1 year.
  Pre stimulus peak values (-30 to 0+) will be compared to post stimulus peak values (0+ to 30+).
Peak values for NOL and SCA for age group 5-12 years | Through study completion, an average of 1 year.
  Pre stimulus peak values (-30 to 0+) will be compared to post stimulus peak values (0+ to 30+).
Reaction time NOL and SCA | Through study completion, an average of 1 year.
  Comparison of average reaction time in seconds of NOL and SCA after nociceptive stimuli/event. measured in seconds.
NOL and SCA reaction during locoregional anaesthesia technique | Through study completion, an average of 1 year.
  Pre stimulus peak values (-30 to 0+) will be compared to post stimulus peak values (0+ to 30+) for both NOL and SCA for nociceptive stimuli placed inside area of the skin covered bij locoregional blockade.

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
There are plans to publish the findings and the participants and their caregivers will be informed of this during the informed consent procedure.

REFERENCES:
- [Background] Ledowski T. Objective monitoring of nociception: a review of current commercial solutions. Br J Anaesth. 2019 Aug;123(2):e312-e321. doi: 10.1016/j.bja.2019.03.024. Epub 2019 Apr 30. PMID 31047645
- [Background] Sabourdin N, Constant I. Monitoring of analgesia level during general anesthesia in children. Curr Opin Anaesthesiol. 2022 Jun 1;35(3):367-373. doi: 10.1097/ACO.0000000000001141. PMID 35671026
- [Background] Gan TJ. Poorly controlled postoperative pain: prevalence, consequences, and prevention. J Pain Res. 2017 Sep 25;10:2287-2298. doi: 10.2147/JPR.S144066. eCollection 2017. PMID 29026331
- [Background] Ferland CE, Vega E, Ingelmo PM. Acute pain management in children: challenges and recent improvements. Curr Opin Anaesthesiol. 2018 Jun;31(3):327-332. doi: 10.1097/ACO.0000000000000579. PMID 29432292
- [Background] Ben-Israel N, Kliger M, Zuckerman G, Katz Y, Edry R. Monitoring the nociception level: a multi-parameter approach. J Clin Monit Comput. 2013 Dec;27(6):659-68. doi: 10.1007/s10877-013-9487-9. Epub 2013 Jul 9. PMID 23835792
- [Background] Klein Tank C, Himantono N, van Uitert A, Malagon I. Evaluation of the nociception level index in the pediatric population: An observational feasibility study. Paediatr Anaesth. 2023 Jun;33(6):495-496. doi: 10.1111/pan.14632. Epub 2023 Jan 22. No abstract available. PMID 36645161
- [Background] Storm H. Changes in skin conductance as a tool to monitor nociceptive stimulation and pain. Curr Opin Anaesthesiol. 2008 Dec;21(6):796-804. doi: 10.1097/ACO.0b013e3283183fe4. PMID 18997532
- [Background] Chemam S, Cailliau E, Bert D, Tavernier B, Constant I, Sabourdin N. Nociception level response to calibrated stimulations in children: First assessment of the nociception level index in pediatric anesthesia. Anaesth Crit Care Pain Med. 2023 Jun;42(3):101207. doi: 10.1016/j.accpm.2023.101207. Epub 2023 Mar 1. PMID 36863410
- [Background] Storm H. Skin conductance and the stress response from heel stick in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2000 Sep;83(2):F143-7. doi: 10.1136/fn.83.2.f143. PMID 10952711
- [Background] Harrison D, Boyce S, Loughnan P, Dargaville P, Storm H, Johnston L. Skin conductance as a measure of pain and stress in hospitalised infants. Early Hum Dev. 2006 Sep;82(9):603-8. doi: 10.1016/j.earlhumdev.2005.12.008. Epub 2006 Feb 28. PMID 16507342
- [Background] Walas W, Halaba Z, Kubiaczyk A, Piotrowski A, Latka-Grot J, Szczapa T, Romul M, Maroszynska I, Malinowska E, Rutkowska M, Skrzypek M, Smigiel R. Skin conductance measurement for the assessment of analgosedation adequacy in infants treated with mechanical ventilation: A multicenter pilot study. Adv Clin Exp Med. 2020 Sep;29(9):1117-1121. doi: 10.17219/acem/126286. PMID 32937040
- [Background] Karpe J, Misiolek A, Daszkiewicz A, Misiolek H. Objective assessment of pain-related stress in mechanically ventilated newborns based on skin conductance fluctuations. Anaesthesiol Intensive Ther. 2013 Jul-Sep;45(3):134-7. doi: 10.5603/AIT.2013.0028. PMID 24092508
- [Background] Sabourdin N, Arnaout M, Louvet N, Guye ML, Piana F, Constant I. Pain monitoring in anesthetized children: first assessment of skin conductance and analgesia-nociception index at different infusion rates of remifentanil. Paediatr Anaesth. 2013 Feb;23(2):149-55. doi: 10.1111/pan.12071. Epub 2012 Nov 21. PMID 23170802
- [Background] Storm H. "Pain monitoring in anesthetized children: first assessment of skin conductance and analgesia-nociception index at different infusion rates of remifentanil", recommended preset values for the skin conductance equipment was not used. Paediatr Anaesth. 2013 Aug;23(8):761-3. doi: 10.1111/pan.12203. No abstract available. PMID 23822183
- [Background] Ledowski T, Paech MJ, Storm H, Jones R, Schug SA. Skin conductance monitoring compared with bispectral index monitoring to assess emergence from general anaesthesia using sevoflurane and remifentanil. Br J Anaesth. 2006 Aug;97(2):187-91. doi: 10.1093/bja/ael119. Epub 2006 May 23. PMID 16720673
- [Background] Ledowski T, Bromilow J, Paech MJ, Storm H, Hacking R, Schug SA. Skin conductance monitoring compared with Bispectral Index to assess emergence from total i.v. anaesthesia using propofol and remifentanil. Br J Anaesth. 2006 Dec;97(6):817-21. doi: 10.1093/bja/ael278. Epub 2006 Oct 22. PMID 17060330
- [Background] Davidson A, Skowno J. Neuromonitoring in paediatric anaesthesia. Curr Opin Anaesthesiol. 2019 Jun;32(3):370-376. doi: 10.1097/ACO.0000000000000732. PMID 30893116
- [Background] Wang F, Zhang J, Yu J, Tian M, Cui X, Wu A. Variation of bispectral index in children aged 1-12 years under propofol anesthesia: an observational study. BMC Anesthesiol. 2019 Aug 7;19(1):145. doi: 10.1186/s12871-019-0815-6. PMID 31390975
- [Background] Ziesenitz VC, Vaughns JD, Koch G, Mikus G, van den Anker JN. Pharmacokinetics of Fentanyl and Its Derivatives in Children: A Comprehensive Review. Clin Pharmacokinet. 2018 Feb;57(2):125-149. doi: 10.1007/s40262-017-0569-6. PMID 28688027
- [Background] Edry R, Recea V, Dikust Y, Sessler DI. Preliminary Intraoperative Validation of the Nociception Level Index: A Noninvasive Nociception Monitor. Anesthesiology. 2016 Jul;125(1):193-203. doi: 10.1097/ALN.0000000000001130. PMID 27171828